**Unique Protocol ID: 2025/284** 

Brief Title: Effect of Foot Bath on Pain, Sleep, and Comfort Levels After Abdominal Surgery

Official Title: Effect of Foot Bath on Pain, Sleep, and Comfort Levels After Abdominal Surgery:

A Randomized Controlled Trial

25.08.2025

EFFECT OF FOOT BATH ON PAIN, SLEEP, AND COMFORT LEVELS AFTER

ABDOMINAL SURGERY: A RANDOMISED CONTROLLED STUDY

MATERIALS AND METHODS

Data Evaluation

Descriptive statistics (mean ± standard deviation, median, first and third quartiles, number (n), and

percentages (%) for categorical outcomes) and inferential statistics will be used. The Kolmogorov

Smirnov test will be used to determine whether the data are normally distributed. For normally

distributed data, parametric tests (ANOVA, t-test, etc.) will be used for intergroup comparisons. For

non-normally distributed data, nonparametric analysis methods (Mann Whitney U test, Kruskal Wallis

test) will be used for intergroup comparisons. If statistical significance is detected in the Kruskal Wallis

test, which tests three or more variables, the Bonferroni-corrected Mann Whitney U test will be used to

find the reason for the difference. For within-group comparisons, ANOVA (for normally distributed

data) or the Friedman test (for data not showing a normal distribution) will be performed. The IBM

SPSS (V. 31.0) software package will be used for statistical analyses. The statistical significance

threshold will be set at p < .05.

Data will be collected by a single researcher. Each question on the data collection forms will be directed

to the participant, and the answer will be recorded on the form by the researcher. Therefore, it is

predicted that there will be no or very little (<5%) data loss. "A complete case analysis will be performed,

including only participants with no missing data for the primary outcome variables."

Precautions have been taken against the risk of data loss. "To mitigate the risk of possible sample loss,

it has been decided to include 48 patients in each group."